CLINICAL TRIAL: NCT06155747
Title: Transmission and Acquisition of Nontuberculous Mycobacteria Outbreak Investigation (TrANsMIt)
Acronym: C
Status: Recruiting | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-4062
Record Dates: First submitted 2023-05-05; First posted 2023-12-04 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Nontuberculous Mycobacterial Pulmonary Infection; Outbreak Investigation; Healthcare Associated Infection; Mycobacterium Infections
Keywords: Epidemiology; Nontuberculous Mycobacterial Pulmonary Infection; Outbreak investigation; Healthcare Associated Infection; Infection transmission; Infection acquisition
MeSH Terms: conditions — Cross Infection; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole genome sequenced nontuberculous mycobacteria isolates will be retained in the National Jewish Health biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People infected with related NTM isolates identified as having membership in a related cluster: Characterize the source(s) of acquisition and/or direct or indirect patient-to-patient transmission of NTM within a healthcare setting among participants with highly related isolates.
  Interventions: Other: Epidemiologic investigation

INTERVENTIONS:
Other: Epidemiologic investigation — Identification of:
  1. overlaps in source(s) of care between participants with NTM isolates in a healthcare center.
  2. environmental NTM isolates that are highly related to respiratory isolates.
  3. common water source exposure among subjects with clustered NTM infections via shared home of residence watershed.

SUMMARY:
The goal of this observational study is to facilitate standardized nontuberculous mycobacteria (NTM) outbreak investigations in healthcare centers. The main questions it aims to answer are:

* Are respiratory NTM isolates identified as having membership in a suspected healthcare outbreak highly related based on whole genome sequencing?
* Does epidemiologic investigation support healthcare-associated patient-to-patient NTM transmission?
* Does healthcare environmental sampling support healthcare-associated NTM acquisition? If healthcare-associated NTM outbreaks are suspected, participants identified as having membership in a cluster of highly-related NTM infections will complete a demographic questionnaire.

DETAILED DESCRIPTION:
This study is a parallel multi-site study of people cared for in a healthcare center who are identified with highly similar respiratory nontuberculous mycobacteria (NTM) isolates. The Advanced Diagnostic Laboratories (ADx) biorepository collects non-standardized, voluntarily submitted respiratory isolates from healthcare centers throughout the U.S. for the purpose of culture, molecular identification, and WGS. The Transmission and Acquisition of Nontuberculous Mycobacteria Outbreak Investigation (TrANsMIt) study is designed to provide resources to systematically collect data to perform an outbreak investigation on people in a suspected healthcare-associated NTM outbreak. Respiratory NTM isolates will undergo WGS to identify infections that are highly related and falling into clusters in order to determine if the source of NTM infection may be a healthcare-associated outbreak. The investigators integrated clinical and epidemiological research methods to adapt a CDC standardized, and validated Healthcare-Associated Infection Outbreak Investigation Toolkit to retrospectively collect data for suspected healthcare-associated NTM outbreak investigations. Through consultation with subject matter experts and scientific literature review, the investigators modified the CDC Healthcare-Associated Infection Outbreak Investigation Abstraction Form, designed to be utilized in local investigations of common healthcare-associated infections to develop the Healthcare-associated links in transmission of NTM (HALT NTM) study Outbreak Investigation Abstraction Toolkit. The HALT NTM Toolkit is a Health Insurance Portability and Accountability Act (HIPAA) compliant, web-based, branching logic questionnaire that uses integrated clinical and epidemiological research methods to perform an epidemiologic investigation to identify overlaps in space and time with mapping of visits and source(s) of care among patients with highly similar NTM isolates in a Center. Additionally, the Toolkit assesses detailed Center-specific IP&C measures utilized the healthcare system. Utilizing the HALT NTM toolkit, the TrANsMit study facilitates a standardized, stepwise process by which healthcare centers perform an internal epidemiologic evaluation of patients identified as part of an NTM cluster. Since clustered NTM isolates could originate from a shared healthcare source, dust and water biofilms from the healthcare environment are collected. NTM are recovered, identified, and sequenced as described to determine if the respiratory NTM strain genotype is similar to those recovered from the healthcare environment. Through a collaborative agreement, TrANsMIt is available to U.S. healthcare centers to conduct a standardized, independent, confidential NTM outbreak investigation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant of any age who has a history of NTM or a first positive NTM culture collected as part of routine clinical care from expectorated sputum, induced sputum and/or bronchoalveolar lavage.

Exclusion Criteria:

* No NTM respiratory culture

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female participant of any age who has a history of respiratory NTM or a first positive NTM culture collected as part of routine clinical care from expectorated sputum, induced sputum and/or bronchoalveolar lavage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Epidemiologic Investigation | 5 years
  Identification of a shared healthcare-associated source(s) between patients in a healthcare center.
Dust and Water Biofilm Collection | 5 years
  Identification of healthcare dust and water biofilm NTM isolates that are highly related to the isolates recovered from subjects within a healthcare system.
Home of Residence Watershed Mapping | 5 years
  The primary endpoint is identification of common watersheds among subjects infected with clustered NTM isolates.

SECONDARY OUTCOMES:
Epidemiologic Investigation | 5 years
  Incidence and prevalence of CF NTM species/subspecies by geographical region. Between Center comparisons of genetic similarity and patterns of potential transmission.
  Banking of isolates for ex vivo analysis.
Healthcare Environment Dust and Water Biofilm Collection | 5 years
  Incidence and prevalence of healthcare-associated dust and water biofilm NTM species/subspecies by geographical region.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. All IPD will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and any additional supporting information will become available 6 months after publication.
Access Criteria: All IPD will be made available upon request.

REFERENCES:
- [Result] Gross JE, Caceres S, Poch K, Hasan NA, Davidson RM, Epperson LE, Lipner E, Vang C, Honda JR, Strand M, Strong M, Saiman L, Prevots DR, Olivier KN, Nick JA. Healthcare-associated links in transmission of nontuberculous mycobacteria among people with cystic fibrosis (HALT NTM) study: Rationale and study design. PLoS One. 2021 Dec 20;16(12):e0261628. doi: 10.1371/journal.pone.0261628. eCollection 2021. PMID 34929010
- [Result] Gross JE, Caceres S, Poch K, Hasan NA, Jia F, Epperson LE, Lipner E, Vang C, Honda JR, Strand M, Calado Nogueira de Moura V, Daley CL, Strong M, Davidson RM, Nick JA. Investigating Nontuberculous Mycobacteria Transmission at the Colorado Adult Cystic Fibrosis Program. Am J Respir Crit Care Med. 2022 May 1;205(9):1064-1074. doi: 10.1164/rccm.202108-1911OC. PMID 35085056
- [Result] Gross JE, Teneback CC, Sweet JG, Caceres SM, Poch KR, Hasan NA, Jia F, Epperson LE, Lipner EM, Vang CK, Honda JR, Strand MJ, Calado Nogueira de Moura V, Daley CL, Strong M, Davidson RM, Nick JA. Molecular Epidemiologic Investigation of Mycobacterium intracellulare Subspecies chimaera Lung Infections at an Adult Cystic Fibrosis Program. Ann Am Thorac Soc. 2023 May;20(5):677-686. doi: 10.1513/AnnalsATS.202209-779OC. PMID 36656594